CLINICAL TRIAL: NCT04782856
Title: Energy Metabolism in Thyroidectomized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20016169; 1R21DK122310-01A1 (NIH)
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Goiter; Hypothyroidism; Thyroid Cancer
MeSH Terms: conditions — Goiter; Hypothyroidism; Thyroid Neoplasms | interventions — Thyroxine; Triiodothyronine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single therapy (Active Comparator): Levothyroxine (LT4) and placebo (a look-alike inactive substance, a "sugar pill") Patients in the LT4 group will be started at a dose of 1.6 mcg/Kg (52 The VCU Investigational Pharmacy will over-encapsulate LT4 plus placebo, in "AM" and "PM" color coded capsules. Patients will be instructed to take the AM drug first thing in the morning with water only, and to wait at least 30 minutes before taking other medications coffee or breakfast. The PM dose will be taken at least 30 minutes before dinner. Dose adjustments will be performed at the 6-week and 3-month follow up visits by an unblinded endocrinologist (Dr. Yavuz) aiming to achieve and maintain a target TSH within the normal range and within ± 0.5 mcIU/ml from the baseline (pre-surgery) TSH, Doses will be rounded to the nearest available formulation.
  Interventions: Drug: Levothyroxine; Drug: Placebo
- Combination therapy (Experimental): Liothyronine/levothyroxine (LT3/LT4) combination therapy. LT4/LT3 group will have 25 mcg of LT4 substituted with 5 mcg LT3 twice daily, to mimic the average daily T3 production form the thyroid The VCU Investigational Pharmacy will over-encapsulate LT4 plus 5 mcg LT3 in "AM" and "PM" color coded capsules. Patients will be instructed to take the AM drug first thing in the morning with water only, and to wait at least 30 minutes before taking other medications coffee or breakfast. The PM dose will be taken at least 30 minutes before dinner. Dose adjustments will be performed at the 6-week and 3-month follow up visits by an unblinded endocrinologist (Dr. Yavuz) aiming to achieve and maintain a target TSH within the normal range and within ± 0.5 mcIU/ml from the baseline (pre-surgery) TSH, Doses will be rounded to the nearest available formulation. No changes will be made in LT3.
  Interventions: Drug: Levothyroxine; Drug: Liothyronine

INTERVENTIONS:
Drug: Levothyroxine — levothyroxine sodium tablet for oral use
  Other Names: L-Thryroxine
Drug: Liothyronine — Liothyronine sodium tablets for oral use treatment of hypothyroidism
  Other Names: Cytomel
  Arms: Combination therapy
Drug: Placebo — inert sugar tablets for oral use blinding for treatment of hypothyroidism
  Other Names: Dextrose
  Arms: Single therapy

SUMMARY:
The purpose of this research study is to measure the changes in energy metabolism (how the body burns energy), cardiovascular function (heart function), and lipid metabolism (cholesterol break down and building) before and after thyroidectomy (surgical removal of thyroid gland) in response to two approved therapies for hypothyroidism: levothyroxine (LT4) or Liothyronine/levothyroxine (LT3/LT4) combination therapy.

DETAILED DESCRIPTION:
In this study, Levothyroxine (LT4) and placebo (a look-alike inactive substance, a "sugar pill") will be compared to Liothyronine/ Levothyroxine (LT3/LT4) combination therapy.

Levothyroxine LT4 and Liothyronine (LT3) are drugs approved by the U. S. Food and Drug Administration (FDA).

All participants will be required follow VCU Health COVID-19 standard of Care screening procedures.

This study requires approximately five study visits The five-study visits required will be a Screening Visit (outpatient), one Baseline Visit, (inpatient) one Six Week Visit, (outpatient), one Three Month Visit and one Six Month Visit (both inpatient). A COVID-19 test will be done 48 hours (2 days) before each of the three-inpatient visit, Baseline Visit, Three Month and Six Month Visit.

Participants will be asked to:

1. Give permission for the researchers to collect information about their medical history from participants and their medical records five times during the study visits and for 5 years after the study visits.
2. Have a Physical exam done 5 times
3. 24-hour energy expenditure recording in the Whole room indirect calorimeter studies 3 times (inpatient overnight stays: Baseline, Three months, and Six months visits)
4. Study drug will be dispensed three times
5. Have study drug dose adjustments two times
6. Genomic blood draw for DNA one time
7. Have blood drawn five times
8. Have an DXA Scan two times
9. Have an Echocardiogram three times
10. Complete questionnaire three times
11. Have Accelerometers sensors laced 3 times (inpatient overnight stays: Baseline, Three months, and Six months visits)
12. ClearSight (blood pressure monitoring) procedure three times
13. Be randomized to take either Levothyroxine LT4 + placebo group or LevothyroxineLT3/Liothyronine LT4 group from baseline through 6 months

Participation in this study will last up to 6 months after surgery. Approximately 30 total individuals will participate in this study

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for total thyroidectomy
2. TSH at screening >0.045<4.5mlU/m
3. Adult men and women Age ≥18-89 years of age
4. Euthyroid patients with clinical indication for total thyroidectomy
5. Indication to total thyroidectomy for benign goiter or thyroid cancer not requiring suppressive thyroid hormone therapy

Exclusion Criteria:

1. Weight <50 or >150 Kg
2. Graves' disease
3. Use of thyroid hormone therapy or thyroid supplements (at screening) except for multinodular goiter
4. Indication for thyroid hormone suppressive therapy following surgery
5. Uncontrolled arterial hypertension stage 2 or greater (>140/90 mm Hg at screening) while on medication (patients with hypertension controlled by therapy will be allowed to participate).
6. Uncontrolled diabetes (HbA1c > 8.% at screening or Fructosamine > 325 mmol/L)
7. History of cardiovascular disease, congestive heart failure or unstable coronary artery disease (angina, coronary event, or revascularization within 6 months); atrial fibrillation; or ventricular arrhythmia,
8. History of major depression or psychosis
9. Patients who are Pregnant, breastfeeding planned pregnancy within six months from the thyroidectomy
10. Any conditions that in the opinion of the PI may impede the successful completion of the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki M Stamatouli, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Therapy | Combination Therapy
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Therapy | Combination Therapy | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Short Term Change in Weight
Description: Weight will be measured in kilograms using a stadiometer
Time Frame: Baseline to 6 months post surgery
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Single Therapy | Combination Therapy
Number analyzed (Participants) | 7 | 5
Kilogram | 1.7 (3.9) | -0.76 (2.1)

2. Primary Outcome: Energy Expenditure (EE)
Description: 24-hour EE will be measured using the whole room indirect calorimeter (WRIC) technique
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: calorie over 24 hours
Arm/Group | Single Therapy | Combination Therapy
Number analyzed (Participants) | 6 | 5
calorie over 24 hours | -39 (68) | 25 (29)

3. Primary Outcome: Change in Cholesterol
Description: Cholesterol will be measured using a standard lipid panel.
Time Frame: Baseline to 6 months post surgery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Single Therapy | Combination Therapy
Number analyzed (Participants) | 7 | 5
mg/dL | 43 (73) | -35 (52)

4. Other Pre Specified Outcome: Change in Quality of Life
Description: ThyPRO-39, a thyroid specific quality of life instrument, was used to assess a participant's quality of life. ThyPRO-39 interrogates 12 individual domains and a composite on the 0 to 100 scale (0 best). A difference of 5 points corresponds to a small to moderate effect between two treatment arms. This outcome represents the change in score between when taken at baseline and then again at 6 months post surgery. The larger the increase in score, the better the improvement in the participant's quality of life. Each domain and the composite are being reported separately.
Time Frame: Baseline to 6 months post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Therapy | Combination Therapy
Number analyzed (Participants) | 7 | 5
score on a scale
  Composite | 14.3 (28.3) | 45 (64.7)
  Domain: Goiter | 23.8 (36.8) | 45 (38)
  Domain: Hyperthyroid | 12.5 (20.4) | 15 (18.1)
  Domain: Hypothyroid | -2.7 (17.2) | 10 (24)
  Domain: Eye | 13.1 (17.3) | 5 (12.6)
  Domain: Tiredness | 11.2 (19.3) | 36.7 (45.1)
  Domain: Cognitive | 14.3 (15.8) | 33.3 (45.3)
  Domain: Anxiety | 14.3 (19.1) | 41.7 (45.2)
  Domain: Depressivity | 2.3 (11.5) | 30 (42.3)
  Domain: Emotional | 9.5 (18.9) | 40 (41.8)
  Domain: Social life | 9.5 (14) | 25 (34.4)
  Domain: Daily life | 7.14 (13.1) | 38.3 (51.2)
  Domain: Appearance | 9.5 (47.2) | 38.3 (62.8)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were assed through regular investigator assessment, study laboratory testing and data reporting from treating physicians
Arm/Group | Single Therapy | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Therapy (N=7) | Combination Therapy (N=6)
Unexpected TSH Suppression (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT04782856/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT04782856/ICF_000.pdf